CLINICAL TRIAL: NCT07121543
Title: Understanding the Biological Drivers of Cervical Cancer and Side Effects From Radiation Therapy
Brief Title: Biological Drivers of Cervical Cancer and Side Effects From Radiation Therapy
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jyoti Mayadev, MD, Professor, Radiation Medicine and Applied Sciences, University of California, San Diego
Other Study IDs: 811012
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancer
Keywords: Radiotherapy; Cervical cancer; Translational research; Biomarkers
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical cancer biopsies and blood collected longitudinally from participants with cervical cancer before, during and after radiotherapy.
  Vaginal tissue biopsies and blood collected longitudinally from participants with cervical cancer before, during and after radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cervical cancer biopsy: Using tumor biopsies collected before, during, and after radiotherapy, the investigators will:
  1. Evaluate if irradiation alters tissue factor expression in tumors.
  2. Determine the temporal changes of biomarkers in the irradiated tumor immune microenvironment.
  Interventions: Radiation: Brachytherapy
- Vaginal apex biopsy: Using vaginal tissue biopsies collected before, during, and after radiotherapy, the investigators will:
  1. Evaluate if irradiation alters biomarkers of fibrosis in the vaginal tissue.
  2. Determine the temporal changes of inflammatory biomarkers that increases the stenosis molecular cascade in the irradiated tumor immune microenvironment.
  Interventions: Radiation: Brachytherapy

INTERVENTIONS:
Radiation: Brachytherapy — Brachytherapy is a cancer treatment where radioactive sources are placed inside or near the tumor.
  Other Names: Internal radiation therapy

SUMMARY:
The goal of this observational study is to learn more about the biology of cervical cancer in women who receive radiation therapy for this condition. The main question it aims to answer is:

Does radiation therapy alter the expression of tissue factor and other molecules in cervical cancer over time?

Participants already scheduled for radiation therapy for cervical cancer as part of their regular medical care will provide blood and biopsies of cervical cancer or of the upper portion of the vagina before, during, and on the last day of radiation therapy.

DETAILED DESCRIPTION:
The standard of care treatment for locally advanced cervical cancer is a combination of chemotherapy with cisplatin and radiotherapy. Although patients have improved outcomes with chemo-radiotherapy, tumor recurrence can occur. In addition, combining chemotherapy with radiotherapy increases treatment-related side effects. While breakthroughs in radiotherapy and immunotherapy have resulted in targeted cancer care, chemotherapy given with radiotherapy is a non-targeted approach. Better strategies to treat cervical cancer are needed.

In this study, the investigators will use tissue and blood from patients with cervical cancer to perform translational research. This is necessary to discover molecular pathways that could be targeted in the future with novel agents, such as radiotherapy and immunotherapy, for the treatment of women with cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Pathological diagnosis of cervical cancer
* Scheduled to receive brachytherapy for cervical cancer

Exclusion Criteria:

* Pregnancy or lactation
* Inability to provide a tissue sample

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with cervical cancer.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Tissue factor expression in tumors | 8 weeks
  Determine the temporal changes of tissue factor expression in the irradiated tumor immune microenvironment.

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Mayadev, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No